CLINICAL TRIAL: NCT03511651
Title: The Effect of Positive End-Expiratory Pressure on Functional Residual Capacity During Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: KY2018-004-02
Record Dates: First submitted 2018-04-08; First posted 2018-04-30 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Mechanical Ventilation; Acute Respiratory Distress Syndrome; Functional Residual Capacity
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FRC at clinical PEEP level (Other): Measuring FRC at clinical PEEP level
  Interventions: Procedure: PEEP
- FRC at clinical PEEP + 5cmH2O (Experimental): Increasing PEEP to clinical PEEP + 5cmH2O
  Interventions: Procedure: PEEP

INTERVENTIONS:
Procedure: PEEP — Two PEEP levels will be used during mechanical ventilation.

SUMMARY:
Although positive end-expiratory pressure (PEEP) has been widely used in mechanical ventilated patients with acute respiratory distress syndrome (ARDS), how to select the "optimal" PEEP is far from consensus. The application of PEEP may result in beneficial effect by recruiting previously collapsed lung areas, harmful effect by over-distending previously aerated lung areas, or a combination of the both. The net effect of PEEP in a certain patient may depend on the recruitability. Because recruitability varies extremely in ARDS patients and strongly correlates with the response to PEEP, estimation of end-expiratory lung volume (EELV) may be essential for individualized setting of PEEP. Whether the FRC changes at different PEEP levels remains unknown.

DETAILED DESCRIPTION:
Although positive end-expiratory pressure (PEEP) has been widely used in mechanical ventilated patients with acute respiratory distress syndrome (ARDS), how to select the "optimal" PEEP is far from consensus. The application of PEEP may result in beneficial effect by recruiting previously collapsed lung areas, harmful effect by over-distending previously aerated lung areas, or a combination of the both. The net effect of PEEP in a certain patient may depend on the recruitability. Because recruitability varies extremely in ARDS patients and strongly correlates with the response to PEEP, estimation of end-expiratory lung volume (EELV) may be essential for individualized setting of PEEP.

Passive spirometry has long been used to measure the lung recruitment volume (VREC). A prolonged expiration to zero end-expiratory pressure (ZEEP) or airway release maneuver is required and PEEP induced lung volume change above functional residual capacity (FRC) is measured. This technique assumes that FRC does not change at different PEEP levels.

This assumption that PEEP has no effect on FRC can date back to the study of Valta et al in the early 1990s. Using respiratory inductive plethysmography (RIP), they found that in ALI/ARDS patients, after expiring from different PEEP levels to ZEEP, the plethysmography signal returned to the same baseline value. They concluded that FRC does not change with PEEP, and that changes of EELV are attributable only to change in ∆EELV. Ranieri et al arrived at similar conclusions by measuring differences in lung volumes at different PEEP levels using standardized pressure-volume (P-V) curves derived from the ventilator circuit monitors. However, Patroniti et al found an elevation of FRC as increasing of PEEP in patients with ARDS. In this study, FRC was measured with the helium dilution technique, and concluded that neglecting this effect resulted in marked underestimation of VREC. Whether the FRC changes at different PEEP levels remains controversial. The aim of the study is to assess the effect of PEEP on FRC during mechanical ventilation.

ELIGIBILITY:
Inclusion criteria include:

1. Diagnosed with ARDS according to the Berlin Definition;
2. Age 18-80 years;
3. Ventilated with volume-controlled ventilation using constant flow;
4. Deep sedation (RASS -4 to -5) and absence of spontaneous breathing (i.e., no triggering during tidal breaths and no inspiratory effort during a 5-second end-expiratory hold).

Exclusion criteria include:

1. Evidence of active air leak from the lung, including bronchopleural fistula, pneumothorax, pneumomediastinum, or existing chest tube;
2. Chest wall and/or abdominal injuries;
3. Evidence suggesting reduced chest wall compliance, such as existing large pleural effusion, thoracic trauma and intra-abdominal hypertension (i.e., intra-abdominal pressure > 20 mmHg).
4. Presence of pacemaker, defibrillator, and implantable pumps).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
The change of FRC | 1) One hour after using clinical PEEP 2) One hour after using clinical PEEP + 5cmH2O
  EELV measurement by ICU ventilator; PEEP Volume measured through airway release. FRC will be calculated as EELV minus PEEP volume. Correlation between EELV, PEEP volume, FRC at two different PEEP levels are tested by linear regression analysis.

SECONDARY OUTCOMES:
The change of PaO2/FiO2 Ratio | 1) One hour after using clinical PEEP 2) One hour after using clinical PEEP + 5cmH2O
  Obtaining PaO2 according to blood gas analysis, and FiO2 according to the ventilator
The change of regional EELV | 1) One hour after using clinical PEEP 2) One hour after using clinical PEEP + 5cmH2O
  Regional EELV will be measured at clinical PEEP and clinical PEEP +5cmH2O
The change of homogeneity of distribution of tidal volume | 1) One hour after using clinical PEEP 2) One hour after using clinical PEEP + 5cmH2O
  EIT is used to monitoring the homogeneity of distribution of tidal volume that was divided into two contiguous regions of interest (ROI) equally, the dependent and non-dependent area. The ratio of relative distribution of tidal ventilation of two ROI was calculated.
The change of driving Pressure | 1) One hour after using clinical PEEP 2) One hour after using clinical PEEP + 5cmH2O
  The change of driving pressure will be measured.
The change of regional FRC | 1) One hour after using clinical PEEP 2) One hour after using clinical PEEP + 5cmH2O
  Regional FRC will be measured at clinical PEEP and clinical PEEP +5cmH2O
The change of blood pressure | 1) One hour after using clinical PEEP 2) One hour after using clinical PEEP + 5cmH2O
  The change of blood pressure will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Jian-Xin Zhou, Beijing, Beijing Municipality, China